CLINICAL TRIAL: NCT01059370
Title: Autonom Dysrefleksi Ved Rygmarvsskade
Brief Title: Autonomic Dysreflexia in Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2009-0112
Record Dates: First submitted 2010-01-19; First posted 2010-01-29 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Autonomic Dysfunction; Spinal Cord Injured
Keywords: Autonomic dysfunction; Spinal cord injured; Neurogenic bowel; Neurogenic bladder
MeSH Terms: conditions — Primary Dysautonomias; Neurogenic Bowel; Urinary Bladder, Neurogenic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autonomic dysrefleksia (Experimental): Autonomic dysreflexia in SCI when emptying bowels or filling bladder
  Interventions: Procedure: bowel emptying

INTERVENTIONS:
Procedure: bowel emptying — Bowel is emptied using Peristeen® irrigation system one day, by digital stimulation another trial day or filling the bladder with saline water on a third trial day. BP is measured by Finometer Pro®, respiration frequency by BIOPACK and skin conductivity measured by Biopack and nor-epinephrine and epinephrine are measured in plasma three times during each examination.
  Other Names: Peristeen; Finometer Pro

SUMMARY:
Autonomic dysreflexia in high spinal cord-injured can be initiated by a full bladder or bowel, or when trying to empty either. This randomised study aims at evaluating whether irrigation procedure or digital stimulation or evacuation of the rectum is less provocative of autonomic dysreflexia. Participants have their bowels emptied on different days, in the morning fasting. Bladder filling with sterile saline water is evaluated on a third day as a control.

ELIGIBILITY:
Inclusion Criteria:

1. People with a spinal cord injury above th6 and with symptoms of autonomic dysreflexia.
2. At least one year post injury.
3. 18 years or older.
4. Informed consent.

Exclusion Criteria:

1. Usage of prophylactic anti-autonomic dysreflexia medication.
2. Pregnant or breastfeeding.
3. People who is not able to follow the sudy protocol.
4. No former major surgery in the abdomen or pelvic region.
5. No former radiotherapy in the pelvic region.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-12; Primary Completion 2011-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Intervention induces 25 % raise in BP compared to baseline measurements. | Outcome are monitored all through bowel or bladder-procedure at each of three study-days, and compaire to measurements at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Søren Laurberg, Professor, Study Chair — University of Århus
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark